CLINICAL TRIAL: NCT00614991
Title: Steady-State Plasma Amprenavir (APV) and Raltegravir (RTG) Pharmacokinetics After Fosamprenavir (FPV) and Raltegravir (RTG) Are Each Administered Alone Versus in Combination With or Without Ritonavir (RTV) Boosting in Healthy Adult Subjects
Brief Title: An Interaction Study to Assess Drug Levels in Healthy Adult Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Garden State Infectious Disease Associates, PA (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: COL111242
Record Dates: First submitted 2008-02-01; First posted 2008-02-14 (Estimated); Results first posted 2016-01-29 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Healthy
Keywords: Healthy Subjects; Pharmacokinetics study; Pharmacokinetics of medications
MeSH Terms: interventions — Raltegravir Potassium; fosamprenavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Group A (Active Comparator): Period 1-Raltegravir 400mg BID Period 2-Fosamprenavir 1400mg BID Period 3-Fosamprenavir 1400mg BID + Raltegravir 400mg BID
  Interventions: Drug: Raltegravir; Drug: Fosamprenavir
- Group B (Active Comparator): Period 1-Raltegravir 400mg BID Period2-Fosamprenavir 1400mg BID + Raltegravir 400mg BID Period 3-Fosamprenavir 1400mg BID
  Interventions: Drug: Raltegravir; Drug: Fosamprenavir
- Group C (Active Comparator): Period 1-Raltegravir 400mg BID Period 2-Fosamprenavir 700mg BID + Ritonavir 100mg BID Period 3-Fosamprenavir 700mg BID + Ritonavir 100mg BID + Raltegravir 400mg BID
  Interventions: Drug: Raltegravir; Drug: Fosamprenavir; Drug: Ritonavir
- Group D (Active Comparator): Period 1-Raltegravir 400mg BID Period 2-Fosamprenavir 700mg BID + Ritonavir 100mg BID + Raltegravir 400mg BID Period 3-Fosamprenavir 700mg BID + Raltegravir 100mg BID
  Interventions: Drug: Raltegravir; Drug: Fosamprenavir; Drug: Ritonavir
- Group E (Active Comparator): Period 1-Raltegravir 400mg BID Period 2-Fosamprenavir 1400mg QD + Ritonavir 100mg QD Period 3-Fosamprenavir 1400mg QD + Ritonavir 100mg QD + Raltegravir 400mg BID
  Interventions: Drug: Raltegravir; Drug: Fosamprenavir; Drug: Ritonavir
- Group F (Active Comparator): Period 1-Raltegravir 400mg BID Period 2-Fosamprenavir 1400mg QD + Ritonavir 100mg QD + Raltegravir 400mg BID Period 3-Fosamprenavir 1400mg QD + Ritonavir 100mg QD
  Interventions: Drug: Raltegravir; Drug: Fosamprenavir; Drug: Ritonavir

INTERVENTIONS:
Drug: Raltegravir — 400mg BID
  Other Names: Isentress MK-0518
Drug: Fosamprenavir — 1400mg BID, 700 mg BID or 1400 mg QD
  Other Names: Lexiva
Drug: Ritonavir — 100 mg BID or QD
  Other Names: Norvir
  Arms: Group C; Group D; Group E; Group F

SUMMARY:
To date, no study has investigated whether there is a drug interaction between the protease inhibitor fosamprenavir and the integrase inhibitor raltegravir. COL111242 is a randomized, open-label, 6-arm, 3-period, drug interaction study to assess steady-state plasma amprenavir (APV) and raltegravir (RTG) pharmacokinetics in 48 healthy, HIV-negative adults after administration of a 7-day regimen of RTG 400mg twice a day (BID) alone and after 14-day regimens of unboosted fosamprenavir (FPV) 1400mg twice daily (BID), FPV 700mg/Ritonavir (RTV) 100mg BID, or FPV 1400mg/ritonavir (RTV) 100mg once daily (QD) with and without concurrent RTG 400mg BID. Blood samples for drug concentration measurement will be collected over 12 hours at the end of each dosing period. Subjects will undergo a physical examination, complete blood count (CBC) with differential, HIV test, hepatitis B/C test, liver function test, renal function analysis, and lipid panel at screening, and all of these tests, except those for HIV and hepatitis B/C, will be repeated at follow-up post-study. Adverse events and adherence (by pill count and medication diary) will be assessed by the investigator/study personnel at the end of each dosing period

DETAILED DESCRIPTION:
This randomized, open-label, six-arm, three-period drug interaction study will recruit 48 healthy volunteers so as to obtain a minimum of 36 evaluable subjects at a single study center in the U.S. The study will have a screening visit, 3 treatment visits for pharmacokinetics (PK) sampling and a follow-up visit. The screening visit will be conducted within 30 days prior to receiving the first dose. Subjects will then be randomized into 1 of 6 treatment groups as shown below:

Cohort Size Period 1 Period 2 Period 3 Sample Days 1 to 7 Days 1-14 Days 1-14

A 8 RTG 400mg BID FPV 1400mg BID FPV 1400mg BID

* RTG 400mg BID

B 8 RTG 400mg BID FPV 1400mg BID FPV 1400mg BID

* RTG 400mg BID

C 8 RTG 400mg BID FPV 700mg BID FPV 700mg BID

* RTV 100mg BID + RTV 100mg BID
* RTG 400mg BID

D 8 RTG 400mg BID FPV 700mg BID FPV 700mg BID

* RTV 100mg BID + RTV 100mg BID
* RTG 400mg BID

E 8 RTG 400mg BID FPV 1400mg QD FPV 1400mg QD

* RTV 100mg QD + RTV 100mg QD
* RTG 400mg BID

F 8 RTG 400mg BID FPV 1400mg QD FPV 1400mg QD

* RTV 100mg QD + RTV 100mg QD
* RTG 400mg BID

Study subjects will enter the clinic in the morning prior to dosing and remain at the center for 12 hours following each dose. Fourteen to 21 days following completion of the third dosing period, study subjects will return to the clinic for follow-up assessment. The total duration of the study will be approximately 86 days from screening through follow up. Blood samples for drug concentration measurement of amprenavir (APV) and raltegravir (RTG) concentrations will be collected over 12 hours at the end of each dosing period (at 0 [baseline], 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post-dose). Subjects will undergo a physical examination, CBC with differential, HIV test, hepatitis B/C test, liver function test, renal function analysis, and lipid panel at screening, and all of these tests except those for HIV and hepatitis B/C will be repeated at follow-up post-study. Adverse events and adherence (by pill count and medication diary) will be assessed by the investigator/study personnel at the end of each dosing period. Evaluable patients will be required to have adhered to at least 95% of their study drug doses. Plasma APV concentrations will be analyzed using a validated high-performance liquid chromatography method with tandem mass spectrometric detection (HPLC/MS/MS) and plasma RTG concentrations by triple quadruple mass spectrometry. Plasma APV and RTG pharmacokinetic parameters measured will include maximum concentration (Cmax), time to maximum concentration (Tmax), minimum concentration (Cmin), and area under the concentration-time curve (AUC). All these parameters, except Tmax, will be log-transformed before statistical analysis. Analysis of variance, considering treatment as a fixed effect and subject as a random effect will be performed using Statistical Analysis Software (SAS), and assuming a treatment ratio for steady-state APV PK parameters as 1.0, the 90% confidence intervals will be within the range 0.81-1.24.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Adequate renal function (calculated creatinine clearance via Cockcroft and Gault method (CrCl) > 50 mL/min);
* Adequate hepatic function (total bilirubin < 2.5mg/dL; hepatic transaminases < 5x normal);
* Adequate hematologic function (absolute neutrophil count [ANC] > 750 neutrophils/mm^3; platelets > 50,000/mm^3; hematocrit > 25%);
* Non-smoker
* Willingness and ability to adhere to treatment and follow-up procedures;
* The ability to understand and sign a written informed consent form.

Exclusion Criteria:

* They fail to meet the above inclusion criteria
* Have an active infection that required parenteral antibiotics or hospitalization within 2 weeks prior to enrollment
* A history of or documented gastrointestinal diseases that impact drug absorption
* Are receiving medications that are contraindicated or result in significant drug-drug interactions with RTV (including, but not limited to, triazolam, astemizole, ergot medications, cisapride, midazolam, bepridil, or rifampin)
* Have a significant documented sulfa allergy (e.g., Stevens-Johnson Syndrome)
* HIV, Hepatitis B or C positive
* Cigarette/cigar/pipe smokers
* They are pregnant or lactating. All other women of childbearing potential must use effective method(s) of contraception throughout the study participation and for 30 days following the end of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David V Condoluci, DO, Principal Investigator — GSIDA

RESULTS

PARTICIPANT FLOW:
Groups:
- Group B: Period 1-Raltegravir 400mg BID Period 2-Fosamprenavir 1400mg BID + Raltegravir 400mg BID Period 3-Fosamprenavir 1400mg BID
- Group D: Period 1-Raltegravir 400mg BID Period 2-Fosamprenavir 700mg BID + Ritonavir 100mg BID + Raltegravir 400mg BID Period 3-Fosamprenavir 700mg BID + Ritonavir 100mg BID
- Group E: Period 1-Raltegravir 400mg BID Period 2-Fosamprenavir 1400mg once daily (QD) + Ritonavir 100mg QD Period 3-Fosamprenavir 1400mg QD + Ritonavir 100mg QD + Raltegravir 400mg BID
Period: Overall Study
Arm/Group | Group A | Group B | Group C | Group D | Group E | Group F
Started | 8 | 9 | 7 | 7 | 7 | 6
Completed | 5 | 6 | 7 | 7 | 6 | 6
Not Completed | 3 | 3 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 3 | 3 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group D: Period 1-Raltegravir 400mg BID Period 2- Fosamprenavir 700mg BID + Ritonavir 100mg BID + Raltegravir 400mg BID Period 3-Fosamprenavir 700mg BID + Ritonavir 100mg BID
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Group D | Group E | Group F | Total
Number analyzed (Participants) | 5 | 6 | 7 | 7 | 6 | 6 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 6 | 6 | 7 | 6 | 6 | 36
  >=65 years | 0 | 0 | 1 | 0 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 5 | 3 | 4 | 2 | 20
  Male | 3 | 2 | 2 | 4 | 2 | 4 | 17
Region of Enrollment [Number; unit: participants]
  United States | 5 | 6 | 7 | 7 | 6 | 6 | 37

OUTCOME MEASURES:

1. Primary Outcome: Cmin/Cmax: Steady-state Plasma Amprenavir (APV) Pharmacokinetics (PK) Following Admin of Fosamprenavir (FPV) 1400mg BID, FPV 700mg/Ritonavir (RTV) 100 mg BID, or FPV 1400mg/RTV 100mg QD With and Without Concurrent Raltegravir (RTG) 400mg BID.
Description: APV minimum concentration (Cmin), maximum concentration (Cmax), area under the plasma concentration-time curve (AUC), and oral clearance (CL/F) as determined from APV concentrations observed in blood samples obtained at baseline, and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours during the BID regimens (FPV 1400mg BID, FPV 700mg/RTV 100 mg BID), and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 24 hours during the QD regimen (FPV 1400mg/RTV 100mg QD). As Groups A and B received the same regimens (albeit in different order), PK data for these two groups were collated, then assessed. For the same reason, PK data from Groups C and D regimens were collated before assessment, as were the PK data from Groups E and F
Time Frame: Day 14 of the FPV 1400mg BID, FPV 1400mg/RAL 400mg BID, FPV 700mg/RTV 100mg BID, FPV 700mg/RTV 100mg/RAL 400mg BID, FPV 1400mg/RTV 100mg QD, and FPV 1400mg/RTV 100mg QD plus RAL 400mg BID regimens
Measure: Mean (90% Confidence Interval); unit: ng/mL
Groups:
- Group A & B: Group A Period 1-Raltegravir 400mg BID Period 2-Fosamprenavir 1400mg BID Period 3-Fosamprenavir 1400mg BID + Raltegravir 400mg BID
  Group B Period 1-Raltegravir 400mg BID Period 2-Fosamprenavir 1400mg BID + Raltegravir 400mg BID Period 3-Fosamprenavir 1400mg BID
- Group C & D: Group C Period 1-Raltegravir 400mg BID Period 2-Fosamprenavir 700mg BID + Ritonavir 100mg BID Period 3-Fosamprenavir 700mg BID + Ritonavir 100mg BID + Raltegravir 400mg BID
  Group D Period 1-Raltegravir 400mg BID Period 2-Fosamprenavir 700mg BID + Ritonavir 100mg BID + Raltegravir 400mg BID Period 3-Fosamprenavir 700mg BID + Ritonavir 100mg BID
- Group E & F: Group E Period 1-Raltegravir 400mg BID Period 2-Fosamprenavir 1400mg QD + Ritonavir 100mg QD Period 3-Fosamprenavir 1400mg QD + Ritonavir 100mg QD + Raltegravir 400mg BID
  Group F Period 1-Raltegravir 400mg BID Period 2-Fosamprenavir 1400mg QD + Ritonavir 100mg QD + Raltegravir 400mg BID Period 3-Fosamprenavir 1400mg QD + Ritonavir 100mg QD
Arm/Group | Group A & B | Group C & D | Group E & F
Number analyzed (Participants) | 11 | 14 | 12
ng/mL
  Cmin (ng/mL) | 0.67 [0.49 to 0.93] | 0.67 [0.50 to 0.90] | 0.83 [0.57 to 1.23]
  Cmax (ng/mL) | 0.83 [0.71 to 0.98] | 0.75 [0.59 to 0.96] | 1.27 [1.02 to 1.58]

2. Secondary Outcome: Number of Participants Who Experienced Adverse Events
Description: Safety/tolerability data included all adverse events (AEs) reported within the time frame of each regimen evaluated. The intent was to compare adverse events for each sequence and not for each regimen. The regimens for which AE information was culled were:
  * RAL 400mg BID alone
  * FPV 1400mg BID alone
  * FPV 700mg/RTV 100 mg BID alone
  * FPV 1400mg/RTV 100mg QD alone
  * FPV 1400mg BID combined with RAL 400mg BID
  * FPV 700mg/RTV 100 mg BID combined with RAL 400mg BID
  * FPV 1400mg/RTV 100mg QD combined with RAL 400mg BID The severity of reported AEs was graded according to DAIDS criteria, Version 1.0 (National Institute of Allergy and Infectious Diseases (NIAID). Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0. Division of Acquired Immunodeficiency Syndrome (DAIDS), Washington D.C.; 2004.
Time Frame: Day 0 through Day 49
Measure: Number; unit: participants
Arm/Group | Group A | Group B | Group C | Group D | Group E | Group F
Number analyzed (Participants) | 5 | 6 | 7 | 7 | 6 | 6
participants | 0 | 4 | 6 | 5 | 5 | 4

3. Primary Outcome: AUC: Steady-state Plasma Amprenavir (APV) Pharmacokinetics (PK) Following Admin of Fosamprenavir (FPV) 1400mg BID, FPV 700mg/Ritonavir (RTV) 100 mg BID, or FPV 1400mg/RTV 100mg QD With and Without Concurrent Raltegravir (RTG) 400mg BID.
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: ng•h/mL
Arm/Group | Group A & B | Group C & D | Group E & F
Number analyzed (Participants) | 11 | 14 | 12
ng•h/mL | 0.81 [0.71 to 0.93] | 0.75 [0.58 to 0.97] | 1.13 [0.95 to 1.35]

4. Primary Outcome: CL/F: Steady-state Plasma Amprenavir (APV) Pharmacokinetics (PK) Following Administration of Fosamprenavir (FPV) 1400mg BID, FPV 700mg/Ritonavir (RTV) 100 mg BID, or FPV 1400mg/RTV 100mg QD With and Without Concurrent Raltegravir (RTG) 400mg BID.
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: L/H
Arm/Group | Group A & B | Group C & D | Group E & F
Number analyzed (Participants) | 11 | 14 | 12
L/H | 1.26 [1.08 to 1.46] | 1.43 [1.08 to 1.89] | 1.05 [0.80 to 1.38]

5. Primary Outcome: Cmin/Cmax: Steady-state Plasma RTG PK Following Admin of FPV 1400mg BID, FPV 700mg/RTV 100 mg BID, or FPV 1400mg/RTV 100mg QD With and Without Concurrent RTG 400mg BID.
Description: RAL minimum concentration (Cmin), maximum concentration (Cmax), area under the plasma concentration-time curve (AUC), and oral clearance (CL/F) as determined from RAL concentrations observed in blood samples obtained at baseline, and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours during the period when RAL 400mg BID was administered with the FPV-Containing BID regimens (FPV 1400mg BID, FPV 700mg/RTV 100 mg BID), and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 24 hours during the period when RAL 400mg BID was administered with the FPV QD regimen (FPV 1400mg/RTV 100mg QD). As Groups A and B received the same regimens (albeit in different order), PK data for these two groups were collated, then assessed. For the same reason, PK data from Groups C and D regimens were collated before assessment, as were the PK data from Groups E and F.
Time Frame: Day 7 of the RAL 400mg BID regimen and Day 14 of the RAL 400mg/FPV 1400mg BID, RAL 400mg/FPV 700mg/RTV 100mg BID, and RAL 400mg BID Plus FPV 1400mg/RTV 100mg QD regimens
Measure: Mean (90% Confidence Interval); unit: ng/mL
Groups:
- Group A & B: Group A Period 1-Raltegravir 400mg BID Period 2-Fosamprenavir 1400mg BID Period 3-Fosamprenavir 1400mg BID + Raltegravir 400mg BID Group B Period 1-Raltegravir 400mg BID Period2-Fosamprenavir 1400mg BID + Raltegravir 400mg BID Period 3-Fosamprenavir 1400mg BID
- Group C & D: Group C Period 1-Raltegravir 400mg BID Period 2-Fosamprenavir 700mg BID + Ritonavir 100mg BID Period 3-Fosamprenavir 700mg BID + Ritonavir 100mg BID + Raltegravir 400mg BID
  Group D Period 1-Raltegravir 400mg BID Period 2-Fosamprenavir 700mg BID + Ritonavir 100mg BID + Raltegravir 400mg BID Period 3-Fosamprenavir 700mg BID + Raltegravir 100mg BID
Arm/Group | Group A & B | Group C & D | Group E & F
Number analyzed (Participants) | 11 | 14 | 12
ng/mL
  Cmin (ng/mL) | 0.32 [0.15 to 0.66] | 0.46 [0.26 to 0.82] | 0.59 [0.27 to 1.30]
  Cmax (ng/mL) | 0.95 [0.64 to 1.43] | 0.44 [0.30 to 0.66] | 0.85 [0.58 to 1.24]

6. Primary Outcome: AUC: Steady-state Plasma Amprenavir (APV) Pharmacokinetics (PK) Following Administration of Fosamprenavir (FPV) 1400mg BID, FPV 700mg/Ritonavir (RTV) 100 mg BID, or FPV 1400mg/RTV 100mg QD With and Without Concurrent Raltegravir (RTG) 400mg BID.
Description: as for outcome 1
Time Frame: as for outcome 5
Measure: Mean (90% Confidence Interval); unit: ng•h/mL
Arm/Group | Group A & B | Group C & D | Group E & F
Number analyzed (Participants) | 11 | 14 | 12
ng•h/mL | 0.71 [0.54 to 0.94] | 0.46 [0.34 to 0.63] | 0.70 [0.52 to 0.94]

7. Primary Outcome: CL/F: Steady-state Plasma Amprenavir (APV) Pharmacokinetics (PK) Following Administration of Fosamprenavir (FPV) 1400mg BID, FPV 700mg/Ritonavir (RTV) 100 mg BID, or FPV 1400mg/RTV 100mg QD With and Without Concurrent Raltegravir (RTG) 400mg BID.
Description: as for outcome 1
Time Frame: as for outcome 5
Measure: Mean (90% Confidence Interval); unit: L/h
Arm/Group | Group A & B | Group C & D | Group E & F
Number analyzed (Participants) | 11 | 14 | 12
L/h | 1.02 [0.88 to 1.19] | 2.30 [1.52 to 3.47] | 1.46 [0.96 to 2.21]

ADVERSE EVENTS:
Time Frame: Reported Adverse Events (AE) included events starting on or after Day 0 through Day 49.
Description: If a subject experienced more than 1 of a given AE, the subject is counted only once for that AE.
Arm/Group | Group A | Group B | Group C | Group D | Group E | Group F
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6 | 0/7 | 0/7 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/5 | 4/6 | 6/7 | 5/7 | 5/6 | 4/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=5) | Group B (N=6) | Group C (N=7) | Group D (N=7) | Group E (N=6) | Group F (N=6)
Nausea/Vomiting/Diarrhea (Gastrointestinal disorders) | 0 | 3 | 5 | 5 | 3 | 3 — cramps/ gas/bloating/heartburn
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 2 | 1 | 0 | 0
Headache (General disorders) | 0 | 0 | 1 | 2 | 0 | 1
Dizzy (General disorders) | 0 | 0 | 1 | 0 | 1 | 1
Dry mouth/loss of appetite (General disorders) | 0 | 0 | 1 | 1 | 1 | 1
Sinus infection/Flu like symptoms (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 (0)
Increased urination (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Numbness of mouth/lips/tongue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sleep disturbance (General disorders) | 0 | 0 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Data for primary outcomes are not available per intervention . Values reported as means are uncertain measure type (data no longer available).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No